

## Study Protocol

Title of Study: Can an adjustable compression garment replace compression bandaging in the treatment of patients with Breast Cancer related upper limb Lymphoedema? A pilot study

Document creation date: March 26<sup>th</sup> 2020

NCT number [not yet assigned]

Identifiers: [NCT ID not yet assigned]



## Study Protocol

**Intervention**: Participants will attend the Physiotherapy Department in Sligo University Hospital for treatment. The will receive Complex decongestive Therapy consisting of 5 Manual Lymphatic drainage treatments, each followed by wrapping with coban compression wrapping (Control Group- standard treatment) or an adjustable compression garment (Experimental Group).

Limb Volume will be measured pre –treatment, after 3 treatments and on the last appointment by a blinded assessor.

All participants will be given advice on exercises, skin care, and weight management.

## Main outcome measure:

Limb Volume measured using the truncated cone formula

**Secondary Outcomes**: Quality of life using Short Form 36 Questionnaire

## **Objectives of Study:**

- 1. Evaluate the effect that an adjustable compression garment has on Lymphoedema volume.
- 2. Explore how this new therapy compares to the current standard treatment
- 3. Identify any adverse effects.